CLINICAL TRIAL: NCT05412849
Title: Is the Radiation Field, Dose and Fractionation Crucial for the Development of Mandibular Complications When Treating Malignancies in the Oropharyngeal Region?
Brief Title: Radiation Field, Dose and Fractionation Related to Mandibular Complications
Status: Recruiting | Type: Observational
Sponsor: Lund University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: LundUH
Record Dates: First submitted 2022-02-08; First posted 2022-06-09 (Actual); Last update posted 2024-05-23 (Actual); Status verified 2024-05

CONDITIONS: Head and Neck Neoplasms; Osteoradionecrosis; Radiotherapy; Complications
MeSH Terms: conditions — Head and Neck Neoplasms; Osteoradionecrosis | interventions — Radiotherapy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Radiation: Radiotherapy — Radiotherapy site, time perspective and dose

SUMMARY:
Radiotherapy is inhibiting the healing capacity of the mandibular bone. Late complications as bone exposure, fracture of the jaw, osteoradionecrosis might be a consequence of this vulnerability. A factor that could be involved in the development of complications is field of radiation. There are limited number of studies investigating this relation.

Retrospective analysis of a head and neck oncology register with prospectively included patients will be performed. Patients will be related to the University hospitals in Lund, Umea, Orebro, Stockholm. A thorough analysis of the medical journals in this group of patients will be performed. Included patients have been treated with combination of surgery and radiotherapy to treat malignancies in the head and neck region. At least 12 months follow up period is needed for inclusion.

The scientific aim is to investigate weather the field of radiation and fractionation is crucial for developing the formentioned complications.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of the head and neck malignancy
* Must have recieved radiotherapy as primary treatment alone or combination treatment together with surgery

Exclusion criteria

* less than 12 months follow up
* Under 18 years of age

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Consecutively included patients treated for head and neck neoplasms with a combination of surgery and radiotherapy.
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Complications related to dose, time and position of radiotherapy | The measurements will be done from the end of radiotherapy and atleast 1 year postoperatively.
  Complications as Osteoradionecrosis will be identified and compared with the dose of radiation, how long ago since the radiotherapy was given and where in the mouth the complication has developed.

CONTACTS AND LOCATIONS:
Overall Officials: Martin Bengtsson, PhD, Principal Investigator — Lund University Hospital
Locations (1):
- Skane University Hospital, Lund, Sweden

IPD SHARING:
Plan to Share IPD: No